CLINICAL TRIAL: NCT06131294
Title: Evaluation of Effectiveness of a Novel Remineralizing Agent: A Randomized Controlled Clinical Trial
Brief Title: Efficacy Evaluation of Two Different Fluoride Applications
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ivoclar Vivadent AG (Industry)
Collaborators: Istanbul Medipol University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LL4470462
Record Dates: First submitted 2023-11-02; First posted 2023-11-14 (Actual); Results first posted 2025-04-20 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-03

CONDITIONS: White Spot Lesion
Keywords: white spot lesion
MeSH Terms: interventions — Fluoride Treatment

STUDY DESIGN:
Intervention Model Description: Split-mouth design: Meaning that each patient receives both treatments, but on different teeth.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Expermental Fluoride Application (Experimental): The two-step system, consisting of Component A (ammonium fluoride solution) and Component B (calcium fluoride application), will be applied once on the white spot lesions one.
  Interventions: Device: Fluoride Application (Experimental Fluoride Application)
- Fluor Protector S (Active Comparator): The ammonium fluoride gel will be applied once on the white spot lesions.
  Interventions: Device: Fluor Protector S

INTERVENTIONS:
Device: Fluoride Application (Experimental Fluoride Application) — Fluoride containing applications are applied on white spot lesions. First solution was air-dried before the second application with the other component was done.
  Arms: Expermental Fluoride Application
Device: Fluor Protector S — Fluor Protector S is applied on white spot lesions.
  Arms: Fluor Protector S

SUMMARY:
The goal of this clinical trial is to evaluate the remineralizing or preservative effect of two different fluoride-containing products. The main question aims to answer how the mineral content of the active white spot lesions change after the treatment with those two fluoride applications in a split-mouth design by measuring their mineral content via QLF technology.

Each patient will receive both treatments in a split-mouth design. It is comparison between an experimental fluoride application and Fluoride Protector S.

ELIGIBILITY:
Inclusion Criteria:

* At least two active non-cavitated white spot lesions on buccal surfaces of anterior teeth or premolars (ICDAS code 1 and 2; Nyvad score 1) in two different quadrants.
* Age between 13 and 50 years
* No untreated caries lesions or periodontal disease
* No systematic disease or medication (such as antidepressants, antibiotics etc.) that affects salivary flow rate
* Subjects claimed regular brushing at least twice a day
* Subjects had to agree to keep the scheduled recall appointments for at least 1 year.

Exclusion Criteria:

* Inactive non-cavitated lesions (Nyvad Score 4)
* Lesions with microcavity, cavitation, chipping or discoloration
* Lesions at buccal side of the molars
* Lesions adjacent to restoration
* Developmental white spot lesions such as enamel hypoplasia
* Pregnancy

Ages: 13 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 23 (Actual)
Dates: Start 2023-02-24 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2024-04-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Burcu Gözetici, Dr., Principal Investigator — Istanbul Medipo University
Locations (1):
- Istanbul Medipo University, Istanbul, Esenler, Turkey (Türkiye)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period took place between February 2023 and May 2023 in the Restorative Dentistry Department of Medipol University Clinic
Units Other Than Participants: Lesions
Period: Overall Study
Arm/Group | Expermental Fluoride Application | Fluor Protector S
Started | 23; 30 Lesions | 23; 30 Lesions
6 month recall | 21; 28 Lesions | 21; 28 Lesions
Completed | 21; 28 Lesions | 21; 28 Lesions
Not Completed | 2; 2 Lesions | 2; 2 Lesions

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Expermental Fluoride Application | Fluor Protector S | Total
Number analyzed (Participants) | 23 | 23 | 46
Age, Customized [Count of Participants; unit: Participants]
  14-40 years old | 23 | 23 | 46
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 18
  Male | 14 | 14 | 28
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Measurement of White Spot Lesions by QLF Parameters: Delta F (Max)
Description: Evaluation of the change in lesion size of white spot areas and mineral content by measurement of QLF parameters:
  - delta F (max) (Percentage of maximal fluorescence loss at lesion sites compared to fluorescence of normal enamel, relative fluorecence loss)
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: percent change (%)
Units Other Than Participants: Lesions
Groups:
- Experimental Fluoride Application: The two-step system, consisting of Component A (ammonium fluoride solution) and Component B (calcium fluoride application), will be applied once on the white spot lesions one.
  Fluoride Application (Experimental Fluoride Application): Fluoride containing applications are applied on white spot lesions. First solution was air-dried before the second application with the other component was done.
Arm/Group | Experimental Fluoride Application | Fluor Protector S
Number analyzed (Participants) | 21 | 21
Number analyzed (Lesions) | 28 | 28
percent change (%) | -28.2 (10.8) | -26.3 (13.2)

2. Primary Outcome: Measurement of White Spot Lesions by QLF Parameters: Delta F (Average)
Description: Evaluation of the change in lesion size of white spot areas and mineral content by measurement of QLF parameters:
  - delta F (average) (Percentage of average fluorescence loss at lesion sites compared to fluorescence of normal enamel, relative fluorecence loss)
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: percent change (%)
Units Other Than Participants: Lesions
Arm/Group | Experimental Fluoride Application | Fluor Protector S
Number analyzed (Participants) | 21 | 21
Number analyzed (Lesions) | 28 | 28
percent change (%) | -12.5 (4.0) | -12.2 (5.4)

3. Primary Outcome: Measurement of White Spot Lesions by QLF Parameters: WSA
Description: Evaluation of the change in lesion size of white spot areas and mineral content by measurement of QLF parameters:
  - white spot area (WSA)
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: WSA in px^2
Units Other Than Participants: Lesions
Arm/Group | Experimental Fluoride Application | Fluor Protector S
Number analyzed (Participants) | 21 | 21
Number analyzed (Lesions) | 28 | 28
WSA in px^2 | 376.0 (404.6) | 361.6 (296.7)

4. Primary Outcome: Measurement of White Spot Lesions by QLF Parameters: Delta Q
Description: Evaluation of the change in lesion size of white spot areas and mineral content by measurement of QLF parameters: delta Q
  - delta Q (fluorescence loss in the lesions times with the area of white spot lesions (delta F x WSA); fluorescence loss is negative per definition as enamal has higher mineral content and thus fluorescence than white spot lesions)
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: delta Q in %px
Units Other Than Participants: Lesions
Arm/Group | Experimental Fluoride Application | Fluor Protector S
Number analyzed (Participants) | 21 | 21
Number analyzed (Lesions) | 28 | 28
delta Q in %px | -6539 (8228) | -5022 (5181)

5. Primary Outcome: Measurement of White Spot Lesions by QLF Parameters: Delta R
Description: Evaluation of the change in lesion size of white spot areas and mineral content by measurement of QLF parameters:
  - delta R (increase of red fluorescence at lesion compared to normal enaml; relative red fluorescence increase)
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: delta R in %
Units Other Than Participants: Lesions
Arm/Group | Experimental Fluoride Application | Fluor Protector S
Number analyzed (Participants) | 21 | 21
Number analyzed (Lesions) | 28 | 28
delta R in % | 26.5 (17.9) | 27.3 (25.5)

6. Primary Outcome: Measurement of White Spot Lesions by QLF Parameters: Delta F (Max)
Description: as for outcome 1
Time Frame: 1 Month
Measure: Mean (Standard Deviation); unit: percent change (%)
Units Other Than Participants: Lesions
Arm/Group | Experimental Fluoride Application | Fluor Protector S
Number analyzed (Participants) | 21 | 21
Number analyzed (Lesions) | 28 | 28
percent change (%) | -26.3 (14.8) | -25.6 (12.2)

7. Primary Outcome: Measurement of White Spot Lesions by QLF Parameters: Delta F (Average)
Description: as for outcome 2
Time Frame: 1 Month
Measure: Mean (Standard Deviation); unit: percent change (%)
Units Other Than Participants: Lesions
Arm/Group | Experimental Fluoride Application | Fluor Protector S
Number analyzed (Participants) | 21 | 21
Number analyzed (Lesions) | 28 | 28
percent change (%) | -12.2 (5.4) | -11.9 (4.7)

8. Primary Outcome: Measurement of White Spot Lesions by QLF Parameters: WSA
Description: as for outcome 3
Time Frame: 1 Month
Measure: Mean (Standard Deviation); unit: WSA in px^2
Units Other Than Participants: Lesions
Arm/Group | Experimental Fluoride Application | Fluor Protector S
Number analyzed (Participants) | 21 | 21
Number analyzed (Lesions) | 28 | 28
WSA in px^2 | 446.8 (493.0) | 444.3 (334.9)

9. Primary Outcome: Measurement of White Spot Lesions by QLF Parameters: Delta Q
Description: as for outcome 4
Time Frame: 1 Month
Measure: Mean (Standard Deviation); unit: delta Q in %px
Units Other Than Participants: Lesions
Arm/Group | Experimental Fluoride Application | Fluor Protector S
Number analyzed (Participants) | 21 | 21
Number analyzed (Lesions) | 28 | 28
delta Q in %px | -7105 (9351) | -6234 (5988)

10. Primary Outcome: Measurement of White Spot Lesions by QLF Parameters: Delta R
Description: as for outcome 5
Time Frame: 1 Month
Measure: Mean (Standard Deviation); unit: delta R in %
Units Other Than Participants: Lesions
Arm/Group | Experimental Fluoride Application | Fluor Protector S
Number analyzed (Participants) | 21 | 21
Number analyzed (Lesions) | 28 | 28
delta R in % | 26.4 (22.7) | 32.7 (20.2)

11. Primary Outcome: Measurement of White Spot Lesions by QLF Parameters: Delta F (Max)
Description: as for outcome 1
Time Frame: 6 Month
Measure: Mean (Standard Deviation); unit: percent change (%)
Units Other Than Participants: Lesions
Arm/Group | Experimental Fluoride Application | Fluor Protector S
Number analyzed (Participants) | 21 | 21
Number analyzed (Lesions) | 28 | 28
percent change (%) | -21.2 (12.0) | -26.1 (13.8)

12. Primary Outcome: Measurement of White Spot Lesions by QLF Parameters: Delta F (Average)
Description: as for outcome 2
Time Frame: 6 Month
Measure: Mean (Standard Deviation); unit: percent change (%)
Units Other Than Participants: Lesions
Arm/Group | Experimental Fluoride Application | Fluor Protector S
Number analyzed (Participants) | 21 | 21
Number analyzed (Lesions) | 28 | 28
percent change (%) | -10.1 (4.9) | -12.5 (5.8)

13. Primary Outcome: Measurement of White Spot Lesions by QLF Parameters: WSA
Description: as for outcome 3
Time Frame: 6 Month
Measure: Mean (Standard Deviation); unit: WSA in px^2
Units Other Than Participants: Lesions
Arm/Group | Experimental Fluoride Application | Fluor Protector S
Number analyzed (Participants) | 21 | 21
Number analyzed (Lesions) | 28 | 28
WSA in px^2 | 238.3 (272.5) | 266.6 (296.3)

14. Primary Outcome: Measurement of White Spot Lesions by QLF Parameters: Delta Q
Description: as for outcome 4
Time Frame: 6 Month
Measure: Mean (Standard Deviation); unit: delta Q in %px
Units Other Than Participants: Lesions
Arm/Group | Experimental Fluoride Application | Fluor Protector S
Number analyzed (Participants) | 21 | 21
Number analyzed (Lesions) | 28 | 28
delta Q in %px | -2628 (3216) | -4181 (5833)

15. Primary Outcome: Measurement of White Spot Lesions by QLF Parameters: Delta R
Description: as for outcome 5
Time Frame: 6 Month
Measure: Mean (Standard Deviation); unit: delta R in %
Units Other Than Participants: Lesions
Arm/Group | Experimental Fluoride Application | Fluor Protector S
Number analyzed (Participants) | 21 | 21
Number analyzed (Lesions) | 28 | 28
delta R in % | 22.4 (17.8) | 29.5 (23.0)

16. Primary Outcome: Measurement of White Spot Lesions by QLF Parameters: Delta F (Max)
Description: as for outcome 1
Time Frame: 12 Month
Measure: Mean (Standard Deviation); unit: percent change (%)
Units Other Than Participants: Lesions
Arm/Group | Experimental Fluoride Application | Fluor Protector S
Number analyzed (Participants) | 21 | 21
Number analyzed (Lesions) | 28 | 28
percent change (%) | -22.6 (12.5) | -25.3 (15.5)

17. Primary Outcome: Measurement of White Spot Lesions by QLF Parameters: Delta F (Average)
Description: as for outcome 2
Time Frame: 12 Month
Measure: Mean (Standard Deviation); unit: percent change (%)
Units Other Than Participants: Lesions
Arm/Group | Experimental Fluoride Application | Fluor Protector S
Number analyzed (Participants) | 21 | 21
Number analyzed (Lesions) | 28 | 28
percent change (%) | -10.5 (5.0) | -11.6 (5.7)

18. Primary Outcome: Measurement of White Spot Lesions by QLF Parameters: WSA
Description: as for outcome 3
Time Frame: 12 Month
Measure: Mean (Standard Deviation); unit: WSA in px^2
Units Other Than Participants: Lesions
Arm/Group | Experimental Fluoride Application | Fluor Protector S
Number analyzed (Participants) | 21 | 21
Number analyzed (Lesions) | 28 | 28
WSA in px^2 | 346.4 (400.7) | 373.5 (345.6)

19. Primary Outcome: Measurement of White Spot Lesions by QLF Parameters: Delta Q
Description: as for outcome 4
Time Frame: 12 Month
Measure: Mean (Standard Deviation); unit: delta Q in %px
Units Other Than Participants: Lesions
Arm/Group | Experimental Fluoride Application | Fluor Protector S
Number analyzed (Participants) | 21 | 21
Number analyzed (Lesions) | 28 | 28
delta Q in %px | -4819 (6078) | -5692 (6400)

20. Primary Outcome: Measurement of White Spot Lesions by QLF Parameters: Delta R
Description: as for outcome 5
Time Frame: 12 Month
Measure: Mean (Standard Deviation); unit: delta R in %
Units Other Than Participants: Lesions
Arm/Group | Experimental Fluoride Application | Fluor Protector S
Number analyzed (Participants) | 21 | 21
Number analyzed (Lesions) | 28 | 28
delta R in % | 20.7 (17.0) | 27.8 (22.3)

21. Secondary Outcome: Severity of White Spot Lesions by ICDAS II Visual Scoring System (Codes)
Description: Evaluation of the clinical status of the lesions:
  0: Sound tooth surface: No evidence of caries after 5 sec air drying
  1. First visual change in enamel: Opacity or discoloration (white or brown) is visible at the entrance to the pit or fissure seen after prolonged air drying
  2. Distinct visual change in enamel visible when wet, lesion must be visible when dry
  3. Localized enamel breakdown (without clinical visual signs of dentinal involvement) seen when wet and after prolonged drying
  4. Underlying dark shadow from dentin
  5. Distinct cavity with visible dentin
  6. Extensive (more than half the surface) distinct cavity with visible dentin
Time Frame: Baseline
Measure: Count of Units; unit: lesions
Units Other Than Participants: lesions
Arm/Group | Experimental Fluoride Application | Fluor Protector S
Number analyzed (Participants) | 21 | 21
Number analyzed (lesions) | 28 | 28
lesions
  ICDAS score 0-1 | 0 | 0
  ICDAS score 2 | 28 | 28
  ICDAS score 3-6 | 0 | 0

22. Secondary Outcome: Severity and Activity of White Spot Lesions by Nyvad Criteria
Description: Evaluation of the clinical status of the lesions:
  0: Sound
  1. Active caries (intact surface)
  2. Active caries (surface discontinuity)
  3. Active caries (cavity)
  4. Inactive caries (intact surface)
  5. Inactive caries (surface discontinuity)
  6. Inactive caries (cavity)
  7. Filling (sound surface)
  8. Filling+active caries
  9. Filling+inactive caries
Time Frame: Baseline
Measure: Count of Units; unit: lesions
Units Other Than Participants: lesions
Arm/Group | Experimental Fluoride Application | Fluor Protector S
Number analyzed (Participants) | 21 | 21
Number analyzed (lesions) | 28 | 28
lesions
  Nyvad score 0 | 0 | 0
  Nyvad score 1 | 28 | 28
  Nyvad score 2-3 | 0 | 0
  Nyvad score 4-6 | 0 | 0
  Nyvad score 7-9 | 0 | 0

23. Secondary Outcome: Severity Transition of White Spot Lesions by ICDAS II Visual Scoring System (Codes)
Description: Evaluation of the clinical status of the lesions:
  * "progression" = ICDAS score increased from 2 to 3
  * "unchanged" = ICDAS score 2
  * "regression" = ICDAS score decreased from 2 to 0 or 1
Time Frame: Baseline to 1 month
Measure: Count of Units; unit: lesions
Units Other Than Participants: lesions
Arm/Group | Experimental Fluoride Application | Fluor Protector S
Number analyzed (Participants) | 21 | 21
Number analyzed (lesions) | 28 | 28
lesions
  "Regression" | 3 | 0
  "Unchanged" | 25 | 27
  "Progression" | 0 | 1

24. Secondary Outcome: Severity and Activity Transition of White Spot Lesions by Nyvad Criteria
Description: Evaluation of the clinical status of the lesions:
  * "progression" = Nyvad score changed from 1 to 2 or 5
  * "unchanged" = Nyvad score 1
  * "regression" = Nyvad score changed from 1 to 0 or 4
Time Frame: Baseline to 1 month
Measure: Count of Units; unit: lesions
Units Other Than Participants: lesions
Arm/Group | Experimental Fluoride Application | Fluor Protector S
Number analyzed (Participants) | 21 | 21
Number analyzed (lesions) | 28 | 28
lesions
  "Regression" | 3 | 0
  "Unchanged" | 25 | 27
  "Progression" | 0 | 1

25. Secondary Outcome: Severity Transition of White Spot Lesions by ICDAS II Visual Scoring System (Codes)
Description: as for outcome 23
Time Frame: Baseline to 6 month
Measure: Count of Units; unit: lesions
Units Other Than Participants: lesions
Arm/Group | Experimental Fluoride Application | Fluor Protector S
Number analyzed (Participants) | 21 | 21
Number analyzed (lesions) | 28 | 28
lesions
  "Regression" | 14 | 4
  "Unchanged" | 14 | 20
  "Progression" | 0 | 4

26. Secondary Outcome: Severity and Activity Transition of White Spot Lesions by Nyvad Criteria
Description: as for outcome 24
Time Frame: Baseline to 6 month
Measure: Count of Units; unit: lesions
Units Other Than Participants: lesions
Arm/Group | Experimental Fluoride Application | Fluor Protector S
Number analyzed (Participants) | 21 | 21
Number analyzed (lesions) | 28 | 28
lesions
  "Regression" | 21 | 14
  "Unchanged" | 7 | 10
  "Progression" | 0 | 4

27. Secondary Outcome: Severity Transition of White Spot Lesions by ICDAS II Visual Scoring System (Codes)
Description: as for outcome 23
Time Frame: Baseline to 12 month
Measure: Count of Units; unit: lesions
Units Other Than Participants: lesions
Arm/Group | Experimental Fluoride Application | Fluor Protector S
Number analyzed (Participants) | 21 | 21
Number analyzed (lesions) | 28 | 28
lesions
  "Regression" | 14 | 7
  "Unchanged" | 13 | 16
  "Progression" | 1 | 5

28. Secondary Outcome: Severity and Activity Transition of White Spot Lesions by Nyvad Criteria
Description: as for outcome 24
Time Frame: Baseline to 12 month
Measure: Count of Units; unit: lesions
Units Other Than Participants: lesions
Arm/Group | Experimental Fluoride Application | Fluor Protector S
Number analyzed (Participants) | 21 | 21
Number analyzed (lesions) | 28 | 28
lesions
  "Regression" | 22 | 12
  "Unchanged" | 5 | 12
  "Progression" | 1 | 4

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Expermental Fluoride Application | Fluor Protector S
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/23
Serious Adverse Events (participants affected / at risk) | 1/23 | 1/23
Other Adverse Events (participants affected / at risk) | 0/23 | 0/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Expermental Fluoride Application (N=23) | Fluor Protector S (N=23)
osteosarcoma (General disorders) | 1 | 1 — One patient had osteosarcoma and was excluded from the study. Osteosarcoma is not related to this clinical study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-21): https://cdn.clinicaltrials.gov/large-docs/94/NCT06131294/Prot_SAP_001.pdf